CLINICAL TRIAL: NCT03570385
Title: Can Diffusion Tensor Imaging (DTI) of the Optic Ways Contributes to Predict the 6 Months Prognosis of Optic Neuritis (ON)?
Acronym: DTI et NOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC17_8828_DTI et NOI
Record Dates: First submitted 2017-11-09; First posted 2018-06-27 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Intervention Model Description: Interventional pilot study with minimal risks and constraints, descriptive, prospective, monocentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Optic Neuritis (Experimental)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI in diffusion tensor (DTI : Diffusion Tensor Imaging)

SUMMARY:
Can diffusion tensor imaging (DTI) of the optic ways contributes to predict the 6 months prognosis of Optic Neuritis (ON)?

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 55 years old
* Clinically suspected optic neuritis defined as a sudden decrease of the visual acuity and/or a damage to the field of vision and/or a defect of the colour vision and/or retro-orbital pain with a relative afferent pupillary defect (except if the optic neuropathy is bilateral or symmetrical), in the absence of a severe retinal macular pathology, and in the absence of a toxic or iatrogenic intake (ethambutol, vfend)
* Clinical optic neuritis duration < 15 days
* First episode of an inflammatory ON
* No corticosteroids in the month before
* Indication to a corticosteroid therapy at high dose to cure the felt symptomatology
* Retinal nerve fibre layer (RNFL) thickness upper 75 µm at initial stage
* Isolated ON, multiple sclerosis or NMO (Neuro Myelitis Optica) - SD (Spectrum Disorder) context
* Having signed informed consent for participating in the study

Exclusion Criteria:

* Contra-indication to MRI

  * Cardiac pacemaker or defibrillator implant
  * Neurosurgical clips
  * Cochlear implants
  * Intra-orbital or encephalic foreign bodies
  * Stents implanted since less than 4 weeks and osteosynthesis equipment implanted since less than 6 weeks
  * Claustrophobia
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty
* Eye examination suggests a pre-existing eye abnormality that could affect the visual function (amblyopia, strong myopia…)
* Pregnant or breastfeeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Study of DTI markers in the assessment of the visual prognosis at 6 months of an inflammatory NO based on RNFL thickness (< ou > 75 µm) | Month 6
  MRI

SECONDARY OUTCOMES:
Study of DTI markers in the assessment of the visual prognosis at 6 months of an inflammatory NO based on visual acuity and/or sensible damage to the field of vision | Month 6
  MRI
Comparison of the structural anomalies detected in DTI to the standard morphological MRI (Coronal T2 Fat-Sat MRI and T1 Gadolinium) for ON | Month 6
  MRI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No